CLINICAL TRIAL: NCT04745000
Title: A Prospective Study to Investigate the Use of Actigraphy as a Novel, Reliable and Non-invasive Study Endpoint to Facilitate Pediatric Pulmonary Arterial Hypertension Trials and Drug Development for Children Ages 0-6 Years
Brief Title: Observational Study of Actigraphy in Pediatric Pulmonary Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Other Study IDs: 20-2341; 75F40119C10090 (Other Grant/Funding Number: FDA_BAA-18-00123)
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Hypertension;Pulmonary;Primary
Keywords: Pediatric; Idiopathic; PAH
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pulmonary Hypertension Participants: Children with Primary Pediatric Pulmonary Arterial Hypertension
- Control Participants: Children with a healthy heart and lungs

SUMMARY:
This study plans to learn more about activity levels in children with pulmonary hypertension. Pulmonary hypertension is a condition where the pressure in the lungs is higher than normal. This can affect the person's heart. The purpose of this study is to see if measuring activity in children with pulmonary hypertension and comparing it to activity in children without pulmonary hypertension can give their doctor helpful information on how they are feeling and how their treatment is working.

ELIGIBILITY:
Inclusion criteria for children with PAH:

1. Ages 0-6 years at the time of consent
2. Current diagnosis of pulmonary hypertension in World Health Organization (WHO) Diagnostic Group 1 as per established clinical criteria including prior catheterization meeting Group 1 criteria
3. Panama Functional Class II-IIIa
4. Must have been receiving an approved oral endothelin receptor antagonist, calcium channel blocker, phosphodiesterase 5 inhibitor, prostanoid and/or soluble guanylate cyclase stimulator for at least 30 days prior to consent, and has been at the current stable dose, other than weight-based adjustments, for at least 30 days prior to consent
5. On stable doses of other medical therapy for 14 days prior to enrollment visit with no dose adjustments, additions, or discontinuations (exception diuretics and anticoagulants; OTC/cold/seasonal allergy medications).

Exclusion criteria for children with PAH:

1. Diagnosis of congenital diaphragmatic hernia, or a chronic lung disease, such as bronchopulmonary dysplasia, or interstitial lung disease
2. Any bone (e.g., osteogenesis imperfecta, ankle, knee, or hip injuries), neuromuscular (e.g., muscular dystrophy), or other pathology that may limit activity (e.g., arthritis)
3. Down syndrome
4. Use of any medications known to limit activity (e.g., sedative)
5. Active infection (may re-screen for enrollment once resolved)
6. Any other cardiovascular, liver, renal, hematologic, gastrointestinal, immunologic, endocrine, metabolic, or central nervous system disease or condition that, in the opinion of the Investigator, may adversely affect the safety of the participant or interfere with the interpretation of study assessments

   Examples:
   1. Current diagnosis of uncontrolled sleep apnea as defined by their physician
   2. Severe renal insufficiency as defined by the requirement for dialysis at screening
   3. Moderate to severe hepatic dysfunction defined as elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) liver function tests, greater than or equal to three times the upper limit of normal at screening
7. Actively listed for transplantation
8. Patient and/or legal guardian has/have an unstable psychiatric condition or is/are mentally incapable of understanding the objectives, nature, or consequences of the trial, or has any condition in which the Investigator's opinion would constitute an unacceptable risk to the participant's safety

Inclusion criteria for control children:

1. Ages 0-6 years at the time of consent
2. In good general health as evidenced by medical history reported by parent/legal guardian during screening and/or available medical records

Exclusion criteria for control children:

1. Known diagnosis of asthma (controlled or uncontrolled)
2. Inability to exercise normally either due to an intellectual disability (e.g., Down Syndrome), or a physical disability which could impede activities of daily living.
3. Child and/or legal guardian has/have an unstable psychiatric condition or is/are mentally incapable of understanding the objectives, nature, or consequences of the trial, or has any condition in which the Investigator's opinion would constitute an unacceptable risk to the participant's safety

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: PH patients of PIs seen in cardiology clinics, and a community sample of healthy control participants
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants Meeting Compliance threshold for wearing actigraphy devices: Visit 1 | Over 14 Days, reported at Day 15 post baseline (Visit 1)
  Actigraphy device wear compliance threshold is a minimum of 4 hours per day, and 8 compliant days out of 14 days of wear time.
Number of Participants Meeting Compliance threshold for wearing actigraphy devices: Visit 2 | Over 14 days, reported at about 6 months post-baseline (Visit 2)
  Actigraphy device wear compliance threshold is a minimum of 4 hours per day, and 8 compliant days out of 14 days of wear time.
Number of skin irritation adverse events: Visit 1 | Over 14 Days, reported at Day 15 post baseline (Visit 1)
Number of skin irritation adverse events: Visit 2 | Over 14 days, reported at about 6 months post-baseline (Visit 2)

SECONDARY OUTCOMES:
Heart rate: Visit 1 | Over 14 Days, reported at Day 15 post baseline (Visit 1)
  Measured via Fitbit.
Heart rate: Visit 2 | Over 14 days, reported at about 6 months post-baseline (Visit 2)
  Measured via Fitbit.
Steps per day: Visit 1 | Over 14 Days, reported at Day 15 post baseline (Visit 1)
  Measured via Fitbit and ActiGraph wGT3x-BT.
Steps per day: Visit 2 | Over 14 days, reported at about 6 months post-baseline (Visit 2)
  Measured via Fitbit and ActiGraph wGT3x-BT.
Miles per day: Visit 1 | Over 14 Days, reported at Day 15 post baseline (Visit 1)
  Measured via Fitbit.
Miles per day: Visit 2 | Over 14 days, reported at about 6 months post-baseline (Visit 2)
  Measured via Fitbit.
Energy expenditure per day (kcal): Visit 1 | Over 14 Days, reported at Day 15 post baseline (Visit 1)
  Measured via Fitbit and ActiGraph wGT3x-BT.
Energy expenditure per day (kcal): Visit 2 | Over 14 days, reported at about 6 months post-baseline (Visit 2)
  Measured via Fitbit and ActiGraph wGT3x-BT.
Active minutes per day: Visit 1 | Over 14 Days, reported at Day 15 post baseline (Visit 1)
  Measured via Fitbit.
Active minutes per day: Visit 2 | Over 14 days, reported at about 6 months post-baseline (Visit 2)
  Measured via Fitbit.
Count of Activity Bouts: Visit 1 | Over 14 Days, reported at Day 15 post baseline (Visit 1)
  Count of Active bouts recorded and defined by the Actigraphy devices.
Count of Activity Bouts: Visit 2 | Over 14 days, reported at about 6 months post-baseline (Visit 2)
  Count of Active bouts recorded and defined by the Actigraphy devices.
Count of Sedentary Bouts: Visit 1 | Over 14 Days, reported at Day 15 post baseline (Visit 1)
  Count of Sedentary Bouts recorded and defined by the Actigraphy devices.
Count of Sedentary Bouts: Visit 2 | Over 14 days, reported at about 6 months post-baseline (Visit 2)
  Count of Sedentary Bouts recorded and defined by the Actigraphy devices.
Activity Count: Visit 1 | Over 14 Days, reported at Day 15 post baseline (Visit 1)
  Count of Activity Events recorded and defined by the Actigraphy devices.
Activity Count: Visit 2 | Over 14 days, reported at about 6 months post-baseline (Visit 2)
  Count of Activity Events recorded and defined by the Actigraphy devices.
Physical Activity intensity: Visit 1 | Over 14 Days, reported at Day 15 post baseline (Visit 1)
  Number of minutes with "Mild", "Moderate", and "Vigorous" physical activity.
Physical Activity intensity: Visit 1 | Over 14 days, reported at about 6 months post-baseline (Visit 2)
  Number of minutes with "Mild", "Moderate", and "Vigorous" physical activity.
Resting oxygen saturation at Baseline | Baseline
Resting oxygen saturation at Visit 2 | About 6 months post baseline
Number of PH Participants with Clinical Worsening (CW) Events | End of Study (Up to 12 months post baseline)
Number of PH Participants with Genetic Mutations or Positive Genetic tests | End of Study (Up to 12 months post baseline)
  Count of PH participants with an observed positive genetic test or genetic mutation.
Natriuretic Peptide Tests - BNP | End of Study (Up to 12 months post baseline)
  Brain natriuretic peptide (BNP): a heart failure marker
Natriuretic Peptide Tests - NT-proBNP) | End of Study (Up to 12 months post baseline)
  N-terminal pro b-type natriuretic peptide (NT-proBNP): a heart failure marker

CONTACTS AND LOCATIONS:
Overall Officials: Dunbar Ivy, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No